CLINICAL TRIAL: NCT00924365
Title: A Natural History Study of HIV Acquired in Infancy or Childhood
Brief Title: Natural History Study of HIV Acquired in Infancy or Childhood
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070087; 07-C-0087
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-04-22

CONDITIONS: HIV Infections
Keywords: Children; AIDS; Toxicity; Development; Puberty; HIV; Pediatrics; HIV Infections
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

SUMMARY:
Background:

* About 10,000 children in the United States have been living with HIV infection since birth. Little is known about the long-term effects of HIV infection and its treatment on the growth and development of these children.
* Because of their disease, many children with HIV face additional difficulties with their health, well-being and development, such as success in school and peer relationships.

Objectives:

* To better understand how HIV infection and the medicines used to treat it affect the growth and development of children, adolescents and young adults who have been infected since birth or when they were very young.
* To develop ways to improve the quality of life for these individuals.

Eligibility:

-HIV-infected patients who were followed by the pediatric HIV program in NCI as of December 2004, or an HIV-infected sibling of a participant.

Design:

* Periodic evaluation of pubertal development; bone mineralization; body composition and fat distribution; liver, kidney and heart status; and behavioral, cognitive and academic or vocational outcome of the study group. Evaluations include the following:
* Physical examinations, including height and weight measurements and skin-fold thickness testing to measure body fat.
* Review of medical records and family history.
* Blood and urine tests, including pregnancy test in females who can bear children.
* DEXA scans (X-ray test to measure bone strength and how much fat, muscle and bone is in the body).
* Neuropsychological testing, including evaluation of language, thinking and problem-solving abilities.
* Magnetic resonance imaging (MRI): Test using a magnetic field and radio waves to examine brain structure and function.
* Oral glucose tolerance test: Blood sampling before and one time after the subject drinks a sugary solution to measure the body's ability to use sugar

DETAILED DESCRIPTION:
Background:

Highly active antiretroviral therapy (HAART) has altered the natural history of HIV disease in children.

The pediatric cohort in this country offers a tremendous opportunity to understand the effect of HIV and ARTs on key developmental and maturational processes.

A thorough understanding of the impact of HIV and ARTs on these long-term processes is extremely relevant as ART programs for HIV-infected children are being developed around the world.

Objective:

To explore the clinical features and impact of HIV infection and antiretroviral therapy in an HIV-infected pediatric cohort.

Eligibility:

Known HIV disease and followed in the NCI pediatric HIV program as of December 2004, or HIV-infected sibling of a participant.

Elgibility for the cardiac sub-study is expanded to include any person with HIV acquired in infancy or young childhood who is older than 7 and meets other inclusion criteria.

Eligibility for cardiac sub-study will also include HIV uninfected subjects (18-30 years of age) who will server as a control group.

Design:

Serial evaluations of pubertal development, bone mineralization, body composition and fat distribution, hepatic, renal, and cardiac status, and behavioral, cognitive, and academic/vocational outcome.

Findings may be shared with the multicenter Pediatric HIV/AIDS Cohort Study and lead to more intensive, focused substudies.

ELIGIBILITY:
* INCLUSION CRITERIA:

Known HIV disease and followed in the NCI pediatric HIV program (on an NCI protocol) as of December 2004, or an HIV-infected sibling of a participant.

Age greater than 6 years.

For children greater than 7 years, ability to give assent if developmentally appropriate.

Receives care from a health care provider not affiliated with the protocol.

INCLUSION CRITERIA FOR CARDIAC IMAGING SUB-STUDY:

HIV positive participants

* Known HIV disease, documented or believed to have been acquired during the first decade of life
* Age greater than 7 years old

HIV negative participants

* HIV negative, documented by a negative ELISA
* Age greater than or equal to 18 years old and less than or equal to 30 years old

EXCLUSION CRITERIA:

Inability or unwillingness to provide informed consent for subjects greater than or equal to 18 years, and inability or unwillingness of one parent/legal guardian to provide consent for subjects less than 18 years.

Clinically significant, systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) which in the judgment of the Principal Investigator would compromise the patient s ability to tolerate this study.

EXCLUSION CRITERIA FOR CARDIAC IMAGING SUB-STUDY:

Subjects with contraindication to MRI scanning. These include but are not limited to the presence of any implanted device that is incompatible with MRI.

Subjects who cannot tolerate an MRI scan or who require sedation for MRI.

Pregnant or lactating women.

History of severe allergic reaction to gadolinium contrast agents.

Estimated glomerular filtration rate less than 60 cc/min/1.73m(2).

Inability or unwillingness to provide informed consent for subjects greater than 18 years, and inability or unwillingness of one parent/legal guardian to provide permission for subjects less than 18 years.

Clinically significant, systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) which in the judgement of the Principanl Investigator (or designee) would compromise the patient s ability to tolerate this study

Some subjects may be excluded from cardiac CT but still eligible to enroll in the rest of the study. Exclusion criteria for the cardiac CT component include:

* Age less than 18 years
* Use of metformin-containing products less than 24 hours prior to contrast administration
* History of Multiple Myeloma

Some subjects may be excluded from receiving contrast but will have a non-contrast cardiac CT. Exclusion from receiving contrast include:

* Cratinine value greater than 1.4 mg/dL
* History of significant allergic reaction to CT contrast agents

Some subjects may receive the cardiac CT but will be excluded from receiving beta-blocker. Exclusion criteria for receiving beta-blocker include:

* Asthma
* Active bronchospasm
* Moderate or severe COPD
* 2nd or 3rd degree AV block
* Decompensated cardiac failure
* Allergy to beta blockers
* Systolic blood pressure less than 100 mm HG
* Resting heart rate at the time of scan less than 60 if regular and less than 65 if irregular

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-02-01; Study Completion 2014-04-22

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Hazra, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gortmaker SL, Hughes M, Cervia J, Brady M, Johnson GM, Seage GR 3rd, Song LY, Dankner WM, Oleske JM; Pediatric AIDS Clinical Trials Group Protocol 219 Team. Effect of combination therapy including protease inhibitors on mortality among children and adolescents infected with HIV-1. N Engl J Med. 2001 Nov 22;345(21):1522-8. doi: 10.1056/NEJMoa011157. PMID 11794218
- [Background] Abrams EJ, Weedon J, Bertolli J, Bornschlegel K, Cervia J, Mendez H, Lambert G, Singh T, Thomas P; New York City Pediatric Surveillance of Disease Consortium. Centers for Disease Control and Prevention. Aging cohort of perinatally human immunodeficiency virus-infected children in New York City. New York City Pediatric Surveillance of Disease Consortium. Pediatr Infect Dis J. 2001 May;20(5):511-7. doi: 10.1097/00006454-200105000-00008. PMID 11368109
- [Background] Belman AL, Ultmann MH, Horoupian D, Novick B, Spiro AJ, Rubinstein A, Kurtzberg D, Cone-Wesson B. Neurological complications in infants and children with acquired immune deficiency syndrome. Ann Neurol. 1985 Nov;18(5):560-6. doi: 10.1002/ana.410180509. PMID 3000281
- [Derived] Unsal AB, Mattingly AS, Jones SE, Purdy JB, Reynolds JC, Kopp JB, Hazra R, Hadigan CM. Effect of Antiretroviral Therapy on Bone and Renal Health in Young Adults Infected With HIV in Early Life. J Clin Endocrinol Metab. 2017 Aug 1;102(8):2896-2904. doi: 10.1210/jc.2017-00197. PMID 28531309
- [Derived] Mattingly AS, Unsal AB, Purdy JB, Gharib AM, Rupert A, Kovacs JA, McAreavey D, Hazra R, Abd-Elmoniem KZ, Hadigan C. T-cell Activation and E-selectin Are Associated With Coronary Plaque in HIV-infected Young Adults. Pediatr Infect Dis J. 2017 Jan;36(1):63-65. doi: 10.1097/INF.0000000000001354. PMID 27749650